CLINICAL TRIAL: NCT05664256
Title: Develop, Implement and Evaluate a Public Food Procurement Policy in Nepal
Brief Title: Evaluation of a Healthy Food Procurement Policy at Municipality-level in Nepal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kathmandu University School of Medical Sciences (Other)
Collaborators: Resolve to Save Lives (Other)
Responsible Party: Principal Investigator, Archana Shrestha, Associate Professor, Kathmandu University School of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 628b9a3dcaeacc9d7bbc90f7
Record Dates: First submitted 2022-11-01; First posted 2022-12-23 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Food Selection
Keywords: Food availability; Healthy Food; Food Procurement Policy
MeSH Terms: conditions — Food Preferences | interventions — Educational Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- policy intervention group (Experimental): The group will receive the policy intervention package.
  Interventions: Other: Build capacity of canteen; Other: Information, Education and Communication materials; Other: Monitoring visit
- policy control group (No Intervention): The group will follow the usual guidelines for food procurement policy at the canteen. After three months, the group will receive the policy intervention package.

INTERVENTIONS:
Other: Build capacity of canteen — The investigators will conduct 1 day orientation training to the school nurse, principal and canteen managers of the facilities.
  Different sessions on basic nutrition concept, healthy eating, healthy cooking practices including purchasing and serving will be conducted.
  The investigators will develop training manuals: training curriculum, facilitators guide, and participants guide, aligning with policy contents.
  Arms: policy intervention group
Other: Information, Education and Communication materials — Posters showing healthy plate model will be displayed on the canteen walls. The fact sheet on healthy eating will be distributed to all the public facilities and make it available at the entrance/ gate of the canteen.
  Arms: policy intervention group
Other: Monitoring visit — A monitoring team from each municipality will be formed. The monitoring plan will be prepared with the team. At least one monitoring visit from the municipality government with onsite feedback will be done.
  Arms: policy intervention group

SUMMARY:
The rise in chronic diseases is attributed to unhealthy eating high in sugar, salt and saturated fats, which is facilitated by the availability and consumption of these unhealthy foods. The investigators will conduct the Randomized Controlled Trial to evaluate the effect of food procurement policy on the food environment in the public facilities like schools, worksites, hospitals, correctional facilities and care homes of four municipalities of Bagmati Province, Nepal. The investigators will develop food procurement policy and get endorsed from each municipality through their legislative process. In three months, the change in the food environment after implementing the policy in public facilities of the respective municipalities will be measured.

DETAILED DESCRIPTION:
Introduction:

Unhealthy foods that are high in sugar, salt and saturated fats significantly contribute to poor population health such as obesity and chronic diseases; and are widely available in public facilities including schools, workplaces and health care facilities. Unhealthy diets are thus influenced by an unhealthy food environment. Today's food environment is dependent on the consumer's choice and is supposed to be challenging. Consumers are not taking healthy choices on their nutrition and health. Thus, promotion of a healthier food environment in public facilities is recognized as the best measure for addressing the adverse health outcomes. Healthy public food procurement consists of procuring, distributing, selling, and/or serving food to facilitate healthier dietary behaviors. The development, implementation and adoption of healthy food procurement policy is regarded as the promising strategy to address the health consequences associated with unhealthy foods. Nepal still is struggling in meeting high standards of safe, nutritious diets for the entire population. Due to the increased market prices of the foods, the purchasing capacity of the country has been affected. There are issues of nutrition transition which have resulted in a lack of dietary diversity. The sales as well as demand of ultra-processed foods are increasing. The typical dietary pattern of refined grains, meat and alcohol is associated with a higher prevalence of overweight and obesity. Deep-fried foods are associated with hypertension; the cereal and vegetable pattern are inversely associated with diabetes prevalence. The foods such as packed foods, canned juices, cold drinks, restaurant foods and other junk foods are sold everywhere which is due to attractive media advertisements; increase in street food, supermarkets, fast food chain industries; quick availability/preparation/consumption; easy carrying and handling with home packing system.

There is sufficient evidence that public food procurement policy with randomized controlled trials (RCTs) shows increasing the consumption and availability of healthy food in public facilities such as school, hospital, correctional facilities and care homes; there is no such study in Nepal. In this study, the investigators will take reference from the World Health Organization Action framework for developing and implementing public food procurement and service policies for a healthy diet. The healthy food procurement and service policy can be a "double duty action" for improving health and reducing all forms of malnutrition in the population. Making public food procurement and service policies healthier is a low-cost strategy that can improve the health and nutritional status, including weight-related outcomes, of the population by increasing the availability and consumption of healthier food in public settings, while simultaneously decreasing availability and consumption of unhealthy food. Different countries have committed to taking action to promote healthy diets and eliminate malnutrition in all its forms, including ensuring healthy food in public facilities.

Rationale:

Unhealthy foods that are high in sugar, salt and saturated fats significantly contribute to poor population health such as obesity and chronic diseases; and are widely available in public facilities including schools, workplaces and health care facilities. People tend to be unaware or ignore the health effects of these unhealthy foods. Improving knowledge on unhealthy eating is necessary but not sufficient to change dietary behaviors at the population level. Therefore, population-level policies and programs are necessary to address unhealthy eating at societal level. Nepal Government recognizes nutrition and food security as a top priority. However, no specific food procurement policy to regulate purchase and availability of healthy foods is in place. Development and implementation of a sustainable public food procurement and service policy will lead to availability of a wider variety of healthier products for the public.

Objectives:

Assess the effectiveness of public food procurement policy implementation.

ELIGIBILITY:
Inclusion Criteria:

Participants inclusion criteria:

* Canteen managers or staff who are directly involved in food procurement and service (purchasing, preparation, serve or sell) at the canteen and available at the time of interview; - Canteen managers or staff age between 15-59 year; and
* who can communicate verbally.

Facilities inclusion criteria:

* facilities: government schools, private schools, government worksites, government hospitals, government care homes and government correctional facilities
* facilities within the surrounding of the selected municipality
* facilities who have their own canteen facilities

Exclusion Criteria:

Participants exclusion criteria

- Voluntarily requesting exclusion from the study

Ages: 15 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 402 (Estimated)
Dates: Start 2023-05-27 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in availability of healthy and unhealthy food options | 3 months
  We will calculate the percentage change in both the availability and sales of the foods such as fruits, vegetables, whole grains, trans fats, high sodium and sugar containing foods.

CONTACTS AND LOCATIONS:
Overall Officials: Archana Shrestha, PHD, Principal Investigator — Associate Professor
Locations (1):
- Budhanilkantha, Hattigauda, Province, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vandevijvere S, Chow CC, Hall KD, Umali E, Swinburn BA. Increased food energy supply as a major driver of the obesity epidemic: a global analysis. Bull World Health Organ. 2015 Jul 1;93(7):446-56. doi: 10.2471/BLT.14.150565. PMID 26170502
- [Background] Influencing food environments for healthy diets. [cited 11 Oct 2022]. Available: https://www.fao.org/policy-support/tools-and-publications/resources-details/en/c/459821/
- [Background] Towards Zero Hunger in Nepal - A Strategic Review of Food Security and Nutrition 2018. In: ReliefWeb [Internet]. [cited 11 Oct 2022]. Available: https://reliefweb.int/report/nepal/towards-zero-hunger-nepal-strategic-review-food-security-and-nutrition-2018
- [Background] Tamrakar D, Shrestha A, Rai A, Karmacharya BM, Malik V, Mattei J, Spiegelman D. Drivers of healthy eating in a workplace in Nepal: a qualitative study. BMJ Open. 2020 Feb 25;10(2):e031404. doi: 10.1136/bmjopen-2019-031404. PMID 32102804
- [Background] Transforming our world: the 2030 Agenda for Sustainable Development. In: UNDP [Internet]. [cited 11 Oct 2022]. Available: https://www.undp.org/ukraine/publications/transforming-our-world-2030-agenda-sustainable-development
- [Background] Amoroso L. The Second International Conference on Nutrition: Implications for Hidden Hunger. World Rev Nutr Diet. 2016;115:142-52. doi: 10.1159/000442100. Epub 2016 May 19. PMID 27197665
- [Background] Diseases N. Global Action Plan for the Prevention and Control of NCDs 2013-2020. World Health Organization; 14 Nov 2013 [cited 11 Oct 2022]. Available: https://www.who.int/publications/i/item/9789241506236
- [Background] Winson A. School Food Environments and the Obesity Issue: Content, Structural Determinants, and Agency in Canadian High Schools. 2008 [cited 11 Oct 2022].
- [Background] Gardner CD, Whitsel LP, Thorndike AN, Marrow MW, Otten JJ, Foster GD, Carson JA, Johnson RK. Food-and-beverage environment and procurement policies for healthier work environments. Nutr Rev. 2014 Jun;72(6):390-410. doi: 10.1111/nure.12116. Epub 2014 May 6. PMID 24801009
- [Background] Dhungana RR, Thapa P, Devkota S, Banik PC, Gurung Y, Mumu SJ, Shayami A, Ali L. Prevalence of cardiovascular disease risk factors: A community-based cross-sectional study in a peri-urban community of Kathmandu, Nepal. Indian Heart J. 2018 Dec;70 Suppl 3(Suppl 3):S20-S27. doi: 10.1016/j.ihj.2018.03.003. Epub 2018 Mar 10. PMID 30595258
- [Background] Healthy Food Systems - Access to Healthy Food and Water. [cited 11 Oct 2022]. Available: https://phasocal.org/alliance-legislative-platform/healthy-food-systems-access-to-healthy-food-and-water/
- [Result] Raine KD, Atkey K, Olstad DL, Ferdinands AR, Beaulieu D, Buhler S, Campbell N, Cook B, L'Abbe M, Lederer A, Mowat D, Maharaj J, Nykiforuk C, Shelley J, Street J. Healthy food procurement and nutrition standards in public facilities: evidence synthesis and consensus policy recommendations. Health Promot Chronic Dis Prev Can. 2018 Jan;38(1):6-17. doi: 10.24095/hpcdp.38.1.03. PMID 29323862
- [Result] Slater J, Green CG, Sevenhuysen G, Edginton B, O'Neil J, Heasman M. The growing Canadian energy gap: more the can than the couch? Public Health Nutr. 2009 Nov;12(11):2216-24. doi: 10.1017/S1368980009990309. Epub 2009 Jun 17. PMID 19531279
- See also: Healthy food procurement and nutrition standards in public facilities: evidence synthesis and consensus policy recommendations. — https://pubmed.ncbi.nlm.nih.gov/29323862/
- See also: Influencing food environments for healthy diets — https://www.fao.org/3/i6484e/i6484e.pdf
- See also: Increased food energy supply as a major driver of the obesity epidemic: a global analysis. — https://pubmed.ncbi.nlm.nih.gov/26170502/
- See also: Towards Zero Hunger in Nepal - A Strategic Review of Food Security and Nutrition 2018. — https://reliefweb.int/report/nepal/towards-zero-hunger-nepal-strategic-review-food-security-and-nutrition-2018
- See also: Drivers of healthy eating in a workplace in Nepal: a qualitative study. — https://pubmed.ncbi.nlm.nih.gov/32102804/
- See also: ransforming our world: the 2030 Agenda for Sustainable Development. — https://sustainabledevelopment.un.org/content/documents/21252030%20Agenda%20for%20Sustainable%20Development%20web.pdf
- See also: The Second International Conference on Nutrition: Implications for Hidden Hunger. — https://pubmed.ncbi.nlm.nih.gov/27197665/
- See also: Global Action Plan for the Prevention and Control of NCDs 2013-2020. — https://www.who.int/publications/i/item/9789241506236
- See also: The growing Canadian energy gap: more the can than the couch? — https://pubmed.ncbi.nlm.nih.gov/19531279/
- See also: Winson A. School Food Environments and the Obesity Issue: Content, Structural Determinants, and Agency in Canadian High Schools. 2008 [cited 11 Oct 2022]. — https://ideas.repec.org/a/spr/agrhuv/v25y2008i4p499-511.html
- See also: Food-and-beverage environment and procurement policies for healthier work environments — https://pubmed.ncbi.nlm.nih.gov/24801009/
- See also: Prevalence of cardiovascular disease risk factors: A community-based cross-sectional study in a peri-urban community of Kathmandu, Nepal — https://pubmed.ncbi.nlm.nih.gov/30595258/
- See also: Healthy Food Systems - Access to Healthy Food and Water Healthy Food Systems — https://phasocal.org/alliance-legislative-platform/healthy-food-systems-access-to-healthy-food-and-water/